CLINICAL TRIAL: NCT04177407
Title: Pelvic Peritoneum Reconstruction Using the Bladder Peritoneum Flap in Laparoscopic Extralevator Abdominoperineal Excision --- A Multi-center, Prospective Single-Arm Cohort Study (IDEAL Phase 2A)
Brief Title: Protocol: Reconstruct the Pelvic Peritoneum Using BPF
Acronym: PPRBPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Director of Department of Gastrointestinal Surgery, West China Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-SA-2019
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: Extralevator abdominoperineal excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective cohort study and fulfill the IDEAL 2A stage principle. Rectal cancer patients undergoing laparoscopic ELAPE, suffering rigid pelvis or huge perineal peritoneum defect, and having difficulty in primary perineal wound closure will be considered eligible. Main exclusion criteria are being complicated with urgent complications, ASA grade > 3 and accompanied with mental illness. Standard laparoscopic ELAPE with pelvic peritoneal floor reconstruction using bladder peritoneum flap are to performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPF group (Experimental): Standard laparoscopic ELAPE with pelvic peritoneal floor reconstruction using bladder peritoneum flap are to performed.
  Interventions: Procedure: Standard laparoscopic ELAPE with pelvic peritoneal floor reconstruction using bladder peritoneum flap are to performed.
- control group (No Intervention): Regarding to the pelvic peritoneum reconstruction, in control group, the pelvic peritoneum will be closed with running suturing. If not possible, the peritoneum covering the surface of the bladder will be secured on the anterior surface of the sacrum with nonabsorbable sutures at the level where the anatomic structure obliterates the pelvic entrance. If neither method was feasible, the pelvic peritoneum defect will be left unclosed.

INTERVENTIONS:
Procedure: Standard laparoscopic ELAPE with pelvic peritoneal floor reconstruction using bladder peritoneum flap are to performed. — Standard laparoscopic ELAPE with pelvic peritoneal floor reconstruction using bladder peritoneum flap are to performed.
  Arms: BPF group

SUMMARY:
Background: Extralevator abdominoperineal excision (ELAPE) may cause various surgical complications including disruption of perineal wound, perineal hernia and adhesive small-bowel obstruction. Pelvic peritoneum reconstruction could prevent those complications, but it may not always be achievable, especially in patients with severe pelvic fibrosis after neoadjuvant radiotherapy. Previous study has reported the application of the pelvic peritoneum reconstruction using the bladder peritoneum flap in laparoscopic ELAPE. The aim of the study is to evaluate the short-term clinical, technical and safety outcomes of pelvic peritoneum reconstruction using the bladder peritoneum flap in laparoscopic ELAPE.

Methods/Design: This is a single -center prospective cohort study and fulfill the IDEAL 2A stage principle. Rectal cancer patients after neoadjuvant radiotherapy and about to undergo laparoscopic ELAPE will be included. Main exclusion criteria are being complicated with urgent complications, ASA grade > 3 and accompanied with mental illness. Patients suffering rigid pelvis or huge perineal peritoneum defect, and having difficulty in primary perineal wound closure will be considered eligible for the baldder peritoneum flap (BPF) group; corresponding rectal cancer patients will be allocated to the control group. After informed consent, 10 patients are planned to be included in the BPF group. Standard laparoscopic ELAPE with pelvic peritoneal floor reconstruction using BPF are to be performed. The surgical safety is to be evaluated after one-year follow-up. Primary endpoints are the occurrence of intraoperative and postoperative complications of pelvic peritoneum reconstruction after ELAPE. Second endpoints are overall complication rate within 30 days after surgery, extent of small intestine falling down to pelvic cavity, and other follow-up consequences within 1 year after surgery.

DETAILED DESCRIPTION:
In rectal cancers, the overall survival will benefit strongly if a negative incisional margin is reached. In order to pursue a negative margin, APR, expecially the extralevator abdominoperineal excision (ELAPE) which introduced by Holm et al had been used to improve the oncological outcome in T3 and T4 rectal cancer. However, ELAPE could bring a gaping hole beyond repair in the pelvic cavity, leading to serious perineal injury and small bowel dropping into pelvic cavity inevitably. Pelvic peritoneal defects can also result in perineal hernia and adhesive small-bowel obstruction (ASBO).

Reconstruction the pelvic peritoneum could prevent the small intestine adhering to the true pelvis by keeping it in the abdominal cavity, thus decrease the occurrence of ASBO and other perineal complications. However, pelvic peritoneum reconstruction may not always be feasible especially in those patients who had received a neoadjuvant radiotherapy and suffered severe tissue fibrosis or those patients who have a large defect of pelvic peritoneum.

Recently the investigators have reported a novel method to reconstruct the pelvic peritoneum under laparoscope in patients with a rigid pelvis. A bladder peritoneum flap was used to cover the defect of pelvic peritoneum. Previous attempts have proved the feasibility of the pelvic peritoneum reconstruction using the bladder peritoneum flap in laparoscopic ELAPE. This protocol is a further study to verify its short-term clinical, technical and safety outcomes.

The objective of this study is to evaluate the short-term clinical, technical and safety outcomes of pelvic peritoneum reconstruction using the bladder peritoneum flap in laparoscopic ELAPE.

This is a multi-center, prospective development study. The method of PPR using the bladder peritoneum flap in laparoscopic ELAPE is at the development stage. And this protocol fulfills the requirement of IDEAL framework stage 2A. Approval of the ethics committee has been obtained from the ethics committee of West China Hospital, Sichuan University (2019 No. 194). The present study was registered on the clinicaltrials.gov. Any technology amendments will be presented to the institutional review board for further assessment. Benefits and risks of the study will be informed to participants. Only participants who signed an informed consent form and agree to participate will be included in this study. Participants have the right to quit the study at any time without any reason. In emergency circumstances, surgeons have the right to end the study. Data of the details will be stored in a database and published after the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 18 to 75.
* ASA grade ≤ 3.
* Pathology confirmed as rectal adenocarcinoma;
* Lower rectal cancer with neoadjuvant (chemo)radiotherapy, and an APR was needed;
* The pelvic peritoneum can't be close by direct suture;
* Patients being able to understand the study protocol and willing to participate in the study, providing written informed consent.

Exclusion Criteria:

* Bladder invaded by tumor or primary bladder cancer.
* severe systemic diseases abibuffecting wound healing (e.g. diabetes, liver cirrhosis or immune compromised status like HIV)
* Sensitivity to anti-adhesion barrier.
* Peritoneal implantation.
* History of severe mental illness.
* Continuous systemic steroid therapy recent 1 month

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
intraoperative complications | within 1 week after surgery.
  Bleeding, flap devitalization, flap laceration, bladder injury and any other event that may cause the failure of the novel method
postoperative complications | 3 month after surgery
  Perineal wound complications and ASBO within 1 year after surgery
postoperative complications | 6 month after surgery
  Perineal wound complications and ASBO within 1 year after surgery
postoperative complications | 12 month after surgery
  Perineal wound complications and ASBO within 1 year after surgery

SECONDARY OUTCOMES:
Overall complication rate within 30 days after surgery. | 30 days after surgery
  Overall complication rate within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holm T, Ljung A, Haggmark T, Jurell G, Lagergren J. Extended abdominoperineal resection with gluteus maximus flap reconstruction of the pelvic floor for rectal cancer. Br J Surg. 2007 Feb;94(2):232-8. doi: 10.1002/bjs.5489. PMID 17143848
- [Background] Yang T, Wei M, Deng X, Meng W, Wang Z. A Novel Laparoscopic Technique With a Bladder Peritoneum Flap Closure for Pelvic Cavity for Patients With Rigid Pelvic Peritoneum After Neoadjuvant Radiotherapy in Laparoscopic Extralevator Abdominoperineal Excision. Dis Colon Rectum. 2019 Sep;62(9):1136-1140. doi: 10.1097/DCR.0000000000001435. PMID 31318767
- [Background] Aggarwal N, Seshadri RA, Arvind A, Jayanand SB. Perineal Wound Complications Following Extralevator Abdominoperineal Excision: Experience of a Regional Cancer Center. Indian J Surg Oncol. 2018 Jun;9(2):211-214. doi: 10.1007/s13193-018-0741-y. Epub 2018 Apr 14. PMID 29887703
- [Background] Butt HZ, Salem MK, Vijaynagar B, Chaudhri S, Singh B. Perineal reconstruction after extra-levator abdominoperineal excision (eLAPE): a systematic review. Int J Colorectal Dis. 2013 Nov;28(11):1459-68. doi: 10.1007/s00384-013-1660-6. Epub 2013 Feb 26. PMID 23440362
- [Background] McCulloch P, Cook JA, Altman DG, Heneghan C, Diener MK; IDEAL Group. IDEAL framework for surgical innovation 1: the idea and development stages. BMJ. 2013 Jun 18;346:f3012. doi: 10.1136/bmj.f3012. PMID 23778427
- [Background] Bengtsson S, Hambraeus A, Laurell G. Wound infections after surgery in a modern operating suite: clinical, bacteriological and epidemiological findings. J Hyg (Lond). 1979 Aug;83(1):41-57. doi: 10.1017/s002217240002581x. PMID 379212
- [Background] Christensen HK, Nerstrom P, Tei T, Laurberg S. Perineal repair after extralevator abdominoperineal excision for low rectal cancer. Dis Colon Rectum. 2011 Jun;54(6):711-7. doi: 10.1007/DCR.0b013e3182163c89. PMID 21552056
- [Derived] Shen Y, Yang T, Deng X, Yang J, Meng W, Wang Z. Pelvic peritoneum reconstruction using the bladder peritoneum flap in laparoscopic extralevator abdominoperineal excision: A multi-center, prospective single-arm cohort study (IDEAL Phase 2A). Medicine (Baltimore). 2020 Jun 19;99(25):e20712. doi: 10.1097/MD.0000000000020712. PMID 32569206